CLINICAL TRIAL: NCT03017573
Title: Prospective Biobanking Study in Cancer Patients Aiming at Better Understand the Link Between the Molecular Alterations of the Tumor Itself, Its Microenvironment and Immune Response (SCANDARE)
Acronym: SCANDARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IC 2016-03
Record Dates: First submitted 2017-01-09; First posted 2017-01-11 (Estimated); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Cancer; Triple-Negative Breast Cancer; Head and Neck Cancer; Cervical Cancer; Sarcoma; Vulva Cancer
Keywords: Immunological biomarkers; molecular profil; Circulating tumor DNA (ctDNA)
MeSH Terms: conditions — Ovarian Neoplasms; Triple Negative Breast Neoplasms; Head and Neck Neoplasms; Uterine Cervical Neoplasms; Sarcoma; Vulvar Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tumor and blood sampling (Experimental): Patients will have a biopsy or a surgery and blood sampling at different time points.
  Interventions: Procedure: Tumor biopsies / Tumor surgery; Procedure: Blood withdrawal

INTERVENTIONS:
Procedure: Tumor biopsies / Tumor surgery — Tumoral tissues samples must be collected at different times points :
  * at the time of surgery
  * before first cycle of adjuvant treatment (if possible)
  * at progression (if possible)
  OR
  * before neoadjuvant therapy
  * at the time of surgery
  * before first cycle of adjuvant treatment (if possible)
  * at progression (if possible)
Procedure: Blood withdrawal — Blood samples must be collected at different times points :
  * at the time of surgery or before the beginning of chemoradiotherapy
  * after surgery or after chemoradiotherapy
  * 6 months after surgery if non recurrence
  * before first cycle of adjuvant treatment or before radiotherapy
  * before second cycle of adjuvant treatment or after radiotherapy
  * at progression
  OR
  * before neoadjuvant therapy
  * during neoadjuvant therapy (post cycle 1)
  * at the time of surgery
  * 6 months after surgery if non recurrence
  * before first cycle of adjuvant treatment or before radiotherapy
  * before second cycle of adjuvant treatment or after radiotherapy
  * at progression

SUMMARY:
SCANDARE is a prospective biobanking study on tumor (+/- nodes), plasma and blood samples at different time points in ovarian, triple negative breast, Head and Neck Cancer, advanced stage treatment-naïve cervical or vulva cancer and sarcoma (breast angiosarcoma and uterine sarcoma) cancers. This study will allowed to identify new molecular and/or immunological biomarkers associated with clinical and biological features of the tumors. All patients will receive standard treatment according to the stage of the diseases and usual procédures.

DETAILED DESCRIPTION:
Patients will have blood and +/- tumor samples at the following times :

1. if eligible for surgery :

   * at surgery (blood + tumor and nodes)
   * after surgery (blood)
   * 6 months after surgery if non recurrence (Blood)
   * before cycle 1 of adjuvant chemotherapy or before radiotherapy (blood + tumor biopsie and nodes if possible)
   * before cycle 2 of adjuvant chemotherapy or after radiotherapy (blood)
   * at progression (blood + tumor biopsie and nodes if possible)
2. if eligible for neoadjuvant chemotherapy :

   * before neoadjuvant therapy (blood + tumor biopsie and nodes)
   * during neoadjuvant therapy (post cycle 1) (blood)
   * at the time of surgery (blood + tumor and nodes)
   * 6 months after surgery if non recurrence (Blood)
   * before cycle 1 of adjuvant chemotherapy or before radiotherapy (blood + tumor biopsie and nodes)
   * before cycle 2 of adjuvant chemotherapy or after radiotherapy (blood)
   * at progression (blood + tumor biopsie and nodes)

ELIGIBILITY:
Inclusion Criteria:

1. Tumor types :

   1. Newly diagnosed treatment-naïve ovarian cancer patients eligible for surgery or neoadjuvant chemotherapy
   2. Newly diagnosed treatment-naïve triple-negative breast cancer patients eligible for surgery or neoadjuvant chemotherapy
   3. Newly diagnosed treatment-naïve head and neck cancer patients eligible for surgery
   4. Newly diagnosed treatment-naïve vulva cancer (all types) or cervical cancer patients with (1) stage Ia - IIa1 with nodal metastasis, postoperative positive margin or parametrial-vaginal involvement, and (2) stage ≥IIa2).
   5. Newly diagnosed treatment-naïve sarcoma cancer patients (1) breast angiosarcoma or (2) uterine sarcoma eligible for surgery or systemic treatment
2. Male or female patients ≥ 18 years of age
3. Signed informed consent

Exclusion Criteria:

1. Male or female patients ≤18 years old
2. Patients with any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
3. Individually deprived of liberty or placed under the authority of a tutor
4. Patients not affiliated to the Social Security System

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050 (Estimated)
Dates: Start 2017-01-06 (Actual); Primary Completion 2029-08-06 (Estimated); Study Completion 2032-01-06 (Estimated)

PRIMARY OUTCOMES:
Correlation between tumor molecular/immunological profile and Baseline clinicobiological features | up to 6 months

SECONDARY OUTCOMES:
Correlation between disease recurrence and molecular and/or immunological biomarkers | up to 24 months
Correlation between genomic alterations and immune parameters | up to 24 months
Correlation between mutations load and immune parameters | up to 24 months
Correlation between ctDNA levels, de novo mutations in ctDNA and immune | up to 24 months
For cervical cancer patient, correlation between ctDNA levels and kinetics, and prognosis, prediction of recurrence | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Edith BORCOMAN, Prof., Principal Investigator — Institut Curie
Locations (6):
- France (6):
  - Institut Bergonie, Bordeaux
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Institut Curie, Paris
  - Institut Curie Hopital Rene Huguenin, Saint-Cloud
  - Institut de Cancérologie de Lorraine - Nancy, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).

REFERENCES:
- [Derived] Hoffmann C, Noel F, Grandclaudon M, Massenet-Regad L, Michea P, Sirven P, Faucheux L, Surun A, Lantz O, Bohec M, Ye J, Guo W, Rochefort J, Klijanienko J, Baulande S, Lecerf C, Kamal M, Le Tourneau C, Guillot-Delost M, Soumelis V. PD-L1 and ICOSL discriminate human Secretory and Helper dendritic cells in cancer, allergy and autoimmunity. Nat Commun. 2022 Apr 13;13(1):1983. doi: 10.1038/s41467-022-29516-w. PMID 35418195